CLINICAL TRIAL: NCT04162535
Title: Contributions to the Elucidation of the Mechanisms and Effects by Which Certain Perianesthetic Interventions Modify Long-term Evolution of Patients With Digestive Cancers Subjected to Surgery
Brief Title: Elucidation of the Mechanisms and Effects of Certain Anesthetic Interventions on Digestive Cancer Patients Subjected to Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Collaborators: Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor (Other); Prof. Dr. I. Chiricuta Institute of Oncology (Other)
Responsible Party: Principal Investigator, Alexandru Alexa, Principal Investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 418/14.11.2018
Record Dates: First submitted 2019-10-13; First posted 2019-11-14 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer
Keywords: Anesthesia; Propofol; Sevoflurane; Lidocaine; Cell Culture
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lidocaine; Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sevoflurane (Experimental): Patients will receive a general volatile anesthesia with Sevoflurane as anesthetic agent
  Interventions: Biological: Blood extraction; Drug: Sevoflurane
- Total intravenous anesthesia (Experimental): Patients will receive a general anesthesia with Propofol as anesthetic agent
  Interventions: Biological: Blood extraction; Drug: Propofol
- Total intravenous anesthesia and Lidocaine (Experimental): Patients will receive a general anesthesia with Propofol as anesthetic agent and will also receive a fully lidocaine infusion according to the lidocaine protocol
  Interventions: Drug: Lidocaine 1% Injectable Solution; Biological: Blood extraction
- Placebo (No Intervention): 10 presumed healthy volunteers that have donated 10 ml of venous blood for serum comparison

INTERVENTIONS:
Drug: Lidocaine 1% Injectable Solution — Lidocaine 1% Injectable Solution Intervention Protocol for the TIVA and Lidocaine Arm
  * Induction: 1.5 mg / kg i.v. bolus before induction (at the vein catch).
  * Maintaining anesthesia: continuous infusion with Lidocaine 2 mg / kg / h, up to a maximum of 200 mg / h during maintenance (after IOT until waking)
  * Infusion with 1% Lidocaine will be reduced to 1.0- 1.5 mg / kg / hour, max 100 mg / hour, for the first 48 hours postop
  Other Names: Antiarrythmic drug
  Arms: Total intravenous anesthesia and Lidocaine
Biological: Blood extraction — The patients will donate after consent 10 ml of blood prior and after surgery for further study
  Other Names: Biologic Human Blood
  Arms: Sevoflurane; Total intravenous anesthesia; Total intravenous anesthesia and Lidocaine
Drug: Sevoflurane — Patients will receive a general volatile anesthesia with Sevoflurane as anesthetic agent
  Other Names: Volatile Anesthetic Drug
  Arms: Sevoflurane
Drug: Propofol — Patients will receive a general anesthesia with Propofol as anesthetic agent
  Other Names: Intravenous Anesthetic Drug
  Arms: Total intravenous anesthesia

SUMMARY:
Digestive cancers (liver, colonic, pancreatic) have a high incidence and high mortality, their population prevalence is also increasing. Given that the anesthesia techniques and the agents used act directly and indirectly on the immune system during the perioperative period, influencing both the treatment and the prognosis of patients with colorectal cancer who undergo elective interventions, a series of perianesthetic interventions have been proposed in order to reduce morbidity-mortality perioperative.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old patients admitted for elective colorectal surgery

Exclusion Criteria:

* Pre-existing chronic pain
* Chronic medication that may interfere with pain: antiepileptics, NSAIDs, corticosteroids
* Contraindications to any of the medications in the study
* Significant psychiatric disorders (Axis I disorder) (major depressive disorders, bipolar disorders, schizophrenia, etc.)
* Hepatic (ALT and / or AST> 2 normal wave) or renal (serum creatinine> 2 mg / dl)
* Convulsive conditions that require medication in the last 2 years
* Planned regional analgesia and / or anesthesia (spinal or epidural)
* Corticosteroid-dependent asthma
* Autoimmune disorders
* Antiarrhythmic drugs (verapamil, propafenone, amiodarone) that may interfere with the antiarrhythmic action of lidocaine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the antiproliferative and apoptotic effects of anesthetic agents | up to 4 years
  The investigators aim to correlate the anticancer effects of two anesthetic techniques with tumor markers (p53;p38) and cell proteins involved in proliferation or apoptosis (IGFR;Bcl-2;Bcl-6).
  The investigators will report if the anesthetic agent used in cancer surgery influences the serologic values of these markers.
Evaluation of patients serum on cell culture | up to 1 week
  The investigators will investigate the serum of the patients who received different types of anesthesia (elective colorectal cancer surgery) by incubating it with colon cell lines (HCT116). The investigators will concentrate on cell proliferation assay.
  The investigators aim to discover how the growth of HCT116 will be influenced by patients' serum in terms of rate of proliferation. The measurements which will be used are Inhibitory Concentration (IC50) measured at 0 , 24 and 48 hours after incubation.
  The concentrations will be measured in mcg/ml.

SECONDARY OUTCOMES:
Lidocaine concentration | up to 4 years
  The investigators aim to determine de plasmatic concentration of lidocaine in the patients serum , which have received lidocaine perioperatively.
  The investigators will do a Mass-Spec analysis of lidocaine
Survival Comparison | up to 5 years
  The investigators will do a follow up for the patients in all the 3 groups. The investigators want to investigate the survival ratio for the patients that had a elective colorectal cancer surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ionescu Daniela, MD PHD DEEA, Study Director — UMF Iuliu Hatieganu Cluj-Napoca
Locations (1):
- Institutu Regional de Gastroenterologie si Hepatologi Prof. Dr. O. Fodor, Cluj-Napoca, Cluj, Romania